CLINICAL TRIAL: NCT00586001
Title: Phase 3 of The Development of A Unified Treatment for Anxiety Disorders
Brief Title: A Unified Treatment for Anxiety Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, David H. Barlow, Professor of Psychology and Psychiatry, Emeritus, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5R34MH070693-02 (NIH)
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Results first posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-11

CONDITIONS: Emotional Disorders; Anxiety Disorders
Keywords: Anxiety; Emotional Disorders; Unified; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Treatment with the Unified Protocol (Arm 1) compared to a 16-week wait list control condition (Arm 2).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Unified Protocol for Transdiagnostic Treatment of Emotional Disorders The UP is a form of transdiagnostic cognitive-behavioral therapy (CBT) for individuals diagnosed with anxiety disorders, depression and related disorders.
  Interventions: Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders
- 2 (No Intervention): Wait-list control: Participants were asked to wait 16 weeks before receiving treatment.

INTERVENTIONS:
Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders — Cognitive-behavioral treatment in development for emotional disorders
  Arms: 1

SUMMARY:
The purpose of this study is to develop a new psychological therapy for a variety of different types of emotional disorders. The study will compare symptoms and functioning of clients who receive the treatment with those who do not, and will include a number of assessments before, during, and after treatment. We predict that patients receiving active treatment will show improved functioning relative to wait-list control.

DETAILED DESCRIPTION:
Emotional disorders, specifically anxiety disorders and depression, are common, chronic, costly, and debilitating to quality of life (Barlow, 2002). Best estimates from various epidemiological studies place the one year prevalence of any anxiety disorder for individuals over 18 at 11.8%, and the one year prevalence of any mood disorder 5.1% (Narrow, Rae, Robins, & Regier, 2002). Lifetime rates are higher. We understand the nature and causes of anxiety and unipolar mood disorders (major depressive disorder and dysthymia) somewhat better than 10 years ago, with evidence pointing to generalized biological and psychological vulnerabilities interacting with specific learning and, sometimes, stressful triggering life events as etiological factors (Barlow, 2002; Brown, Chorpita, & Barlow, 1998). Pharmacological and psychological treatments have been proven effective, at least in the short term, but most studies have ignored the effects of treatment on broad-based patterns of comorbidity that accompany these disorders. Most comorbid disorders are usually additional emotional disorders (Brown, Campbell, Lehman, Grisham, & Mancill, 2001). More importantly, treatment outcomes have been less than satisfactory or ineffective for up to 50% of patients, even for the principal disorder (Nathan & Gorman, 2002). A common pharmacological treatment exists for many emotional disorders, which is selective serotonin re-uptake inhibitors (SSRIs) and closely related compounds. Effective psychological treatments, on the other hand, have been developed to be very specific to each DSM-IV diagnostic category. The purpose of this proposal is to create a unified psychological approach to the emotional disorders. To do, this we will take advantage of recent advances in our understanding of the nature of emotional disorders, as well as emerging knowledge of the process of regulation and change in emotional behavior, in order to distill and refine basic principles of successful psychological treatments. It is expected that this approach will simplify training and dissemination, possibly improve efficacy, and perhaps also shed further light on the nature of emotional disorders. Thus, the specific aims of this proposal are to:

1. Develop and refine a unified psychological treatment for anxiety and non-bipolar mood disorders derived from distilling the major ingredients of current effective approaches in light of advancing knowledge of emotion regulation and modification.
2. Revise and develop methods of evaluating adherence and outcome utilizing this new treatment protocol, focusing not only on symptom reduction but also quality of life and adaptive functioning.
3. Treat a small number of patients with heterogeneous DSM-IV mood and anxiety diagnoses with this new protocol with the purpose of making appropriate modifications for a subsequent pilot study.
4. Conduct a pilot study testing this unified treatment in comparison to a wait-list control condition in order to determine credibility and efficacy in terms of both symptomatic functioning and quality of life, and relating these outcomes to those from more disorder specific treatments.

ELIGIBILITY:
Inclusion Criteria:

* Primary Diagnosis of a DSM-IV Anxiety Disorder

Exclusion Criteria:

* Previous treatment with cognitive-behavioral therapy
* Receiving concurrent psychological treatments during study
* If on psychotropic medicine, requirement for stable dose for at least three months before treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2005-09; Primary Completion 2008-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H Barlow, Ph.D, Principal Investigator — Boston University Center for Anxiety and Related Disorders

REFERENCES:
- [Background] Brown TA, Chorpita BF, Barlow DH. Structural relationships among dimensions of the DSM-IV anxiety and mood disorders and dimensions of negative affect, positive affect, and autonomic arousal. J Abnorm Psychol. 1998 May;107(2):179-92. doi: 10.1037//0021-843x.107.2.179. PMID 9604548
- [Background] Brown TA, Campbell LA, Lehman CL, Grisham JR, Mancill RB. Current and lifetime comorbidity of the DSM-IV anxiety and mood disorders in a large clinical sample. J Abnorm Psychol. 2001 Nov;110(4):585-99. doi: 10.1037//0021-843x.110.4.585. PMID 11727948
- [Background] Barlow DH. Unraveling the mysteries of anxiety and its disorders from the perspective of emotion theory. Am Psychol. 2000 Nov;55(11):1247-63. doi: 10.1037//0003-066x.55.11.1247. PMID 11280938
- [Background] Barlow, D.H., Allen, L., & Choate, M.L. (2006). The Unified Protocol for Treatment of the Emotional Disorders. Unpublished manuscript, Boston University.
- See also: Center for Anxiety and Related Disorders at Boston University webpage — http://www.bu.edu/anxiety

RESULTS

PARTICIPANT FLOW:
Groups:
- Unified Treatment: Unified treatment: The UP is a form of transdiagnostic cognitive-behavioral therapy (CBT) for individuals diagnosed with anxiety disorders, depression and related disorders.
- Wait-List Control: Wait-list control: Participants were asked to wait 16 weeks before receiving treatment.
Period: Overall Study
Arm/Group | Unified Treatment | Wait-List Control
Started | 26 | 11
Completed | 22 | 10
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Unified Treatment | Wait-list Control | Total
Number analyzed (Participants) | 26 | 11 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 11 | 37
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 29.38 [19 to 52] | 30.64 [19 to 43] | 30.01 [19 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 6 | 22
  Male | 10 | 5 | 15
Region of Enrollment [Number; unit: participants]
  United States | 26 | 11 | 37

OUTCOME MEASURES:

1. Primary Outcome: Anxiety Disorders Interview Schedule for DSM-IV
Description: DSM-IV diagnoses of anxiety disorders. Principal and additional diagnoses are assigned a clinical severity rating (CSR) on a scale from 0 (no symptoms) to 8 (extremely severe symptoms), with a rating of 4 or above (definitely disturbing/disabling) passing the clinical threshold for DSM-IV diagnostic criteria.
Time Frame: Measured at pre-treatment (baseline) and post-treatment (month 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unified Treatment | Wait-list Control
Number analyzed (Participants) | 26 | 11
score on a scale
  Pre | 5.23 (0.89) | 5.09 (0.79)
  Post | 3.18 (1.55) | 5.14 (0.80)

2. Secondary Outcome: Structured Interview Guide for the Hamilton Anxiety Rating Scale
Description: Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. Reported scores are the mean total scores.
Time Frame: Measured at pre-treatment (baseline) and post-treatment (month 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unified Treatment | Wait-list Control
Number analyzed (Participants) | 26 | 11
score on a scale
  Pre | 16.15 (7.91) | 14.36 (5.19)
  Post | 7.39 (5.37) | 13.08 (4.22)

3. Secondary Outcome: Structured Interview Guide for the Hamilton Depression Rating Scale
Description: Structured Interview Guide for the Hamilton Depression Rating Scale, items are scored on scale of 0 to 4, higher score meaning a higher severity. Total scores can range from 0 (no symptoms) to 53 (severe). Reported scores are a mean of the total scores.
Time Frame: Measured at pre-treatment (baseline) and post-treatment (month 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unified Treatment | Wait-list Control
Number analyzed (Participants) | 26 | 11
score on a scale
  Pre | 10.35 (5.77) | 10.09 (3.87)
  Post | 5.49 (4.63) | 7.85 (4.01)

4. Secondary Outcome: Positive and Negative Affect Scale
Description: Positive and Negative Affect Schedule-Negative Affectivity; Positive and Negative Affect Schedule-Positive Affectivity; Items are rated on a scale of 1 (very slightly or not at all) to 5 (extremely) relating to how a person feels average feels the indicated emotion. Total scores can range from 20 to 100. Higher scores are more severe. Reported scores are based on mean totals.
Time Frame: Measured at pre-treatment (baseline) and post-treatment (month 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unified Treatment | Wait-list Control
Number analyzed (Participants) | 26 | 11
score on a scale
  Pre; Positive Affect | 28.81 (6.27) | 28.00 (7.19)
  Post; Positive Affect | 32.84 (6.50) | 27.17 (8.61)
  Pre; Negative Affect | 26.62 (5.48) | 24.36 (5.21)
  Post; Negative Affect | 20.57 (4.95) | 22.86 (7.03)

5. Secondary Outcome: Beck Depression Inventory - II
Description: Items are measured on a scale from 0 (little to no symptoms) to 3 (severe). Total scores can range from 0 to 63, higher ratings are more severe. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe. The reported scores are mean total scores.
Time Frame: Measured at pre-treatment (baseline) and post-treatment (month 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unified Treatment | Wait-list Control
Number analyzed (Participants) | 26 | 11
score on a scale
  Pre | 11.96 (7.53) | 11.73 (9.92)
  Post | 4.21 (4.43) | 11.45 (9.64)

6. Secondary Outcome: Beck Anxiety Inventory
Description: Items are scored on a 0 to 3 scale. Total scores range from 0 to 63. 0-9 is minimal, 10-16 is mild, 17-29 is moderate, and 30-63 is severe. Reported scores are a mean of total scores.
Time Frame: Measured at pre-treatment (baseline) and post-treatment (month 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unified Treatment | Wait-list Control
Number analyzed (Participants) | 26 | 11
score on a scale
  Pre | 19.08 (9.93) | 16.91 (6.97)
  Post | 8.27 (6.51) | 12.22 (7.93)

7. Secondary Outcome: Work and Social Adjustment Scale
Description: Items are scored on a 0 to 8 scale. The total score range is 0 to 40. Higher scores are more severe. Reported scores are means of total scores.
Time Frame: Measured at pre-treatment (baseline) and post-treatment (month 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unified Treatment | Wait-list Control
Number analyzed (Participants) | 26 | 11
score on a scale
  Pre | 16.04 (6.53) | 16.46 (2.39)
  Post | 7.62 (5.40) | 13.14 (3.66)

8. Secondary Outcome: Panic Disorder Severity Scale - Self Report Version
Description: Items are rated on a scale of 0 to 4. Scores can range from 0 to 28. Higher scores indicate higher severity of Panic Disorder symptoms
Time Frame: Measured at pre-treatment (baseline) and post-treatment (month 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unified Treatment | Wait-List Control
Number analyzed (Participants) | 26 | 11
score on a scale
  Pre | 7.65 (5.68) | 7.09 (7.04)
  Post | 2.77 (3.01) | 6.20 (7.02)

9. Secondary Outcome: Penn State Worry Questionnaire
Description: The PSWQ is a 16-item questionnaire. Items are rated from 1 to 5, and a total score can range from 16 to 80. Higher scores indicate higher severity of worry symptoms.
Time Frame: Measured at pre-treatment (baseline) and post-treatment (month 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unified Treatment | Wait-List Control
Number analyzed (Participants) | 26 | 11
score on a scale
  Pre | 62.27 (11.54) | 62.55 (10.76)
  Post | 49.18 (13.89) | 60.30 (15.86)

10. Secondary Outcome: Social Interaction Anxiety Scale
Description: The SIAS is a twenty-item measure. Experiences are rated on a 5-point scale from 0 to 4. Experiences are rated on a global period of what is typical. A total score of 60 is possible with cutoffs of 34+ indicative of social phobia and 43+ indicative of social anxiety.
Time Frame: Measured at pre-treatment (baseline) and post-treatment (month 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unified Treatment | Wait-List Control
Number analyzed (Participants) | 26 | 11
score on a scale
  Pre | 28.19 (17.99) | 38.18 (20.03)
  Post | 23.32 (16.76) | 37.60 (20.56)

11. Secondary Outcome: Quality of Life Inventory
Description: The QOLI is a 32 item self-report, asking about the importance of 16 domains of life and a participant's satisfaction in each domain. Scores can range from -48 to 115. Higher scores indicate higher quality of life.
Time Frame: Measured at pre-treatment (baseline) and post-treatment (month 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unified Treatment | Wait-list Control
Number analyzed (Participants) | 26 | 11
score on a scale
  Pre-Treatment | 35.46 (19.52) | 32.45 (10.40)
  Post-Treatment | 46.73 (14.00) | 34.67 (11.15)

12. Secondary Outcome: Yale-Brown Obsessive Compulsive Scale
Description: The Y-BOCS is a 12-item scale used to see symptom severity of obsessions and compulsions. Items are scored from 0 to 4. The total score can range from 0 to 48. A higher score indicates higher symptom severity.
Time Frame: Measured at pre-treatment (baseline) and post-treatment (month 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unified Treatment | Wait-List Control
Number analyzed (Participants) | 26 | 11
score on a scale
  Pre | 8.81 (9.47) | 7.18 (9.91)
  Post | 6.09 (8.17) | 8.65 (8.76)

13. Secondary Outcome: Emotion Regulation Questionnaire - 2
Description: The ERQ-2 is a 16 item self-report. Items are scored from 1 to 7, and focus on emotional experience and emotional expression. Scores can range from 16 to 112, and higher scores indicate stronger cognitive reappraisal and expressive suppression abilities.
Time Frame: Measured at pre-treatment (baseline) and post-treatment (month 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unified Treatment | Wait-list Control
Number analyzed (Participants) | 26 | 11
score on a scale
  Pre-Treatment | 55.40 (16.82) | 60.36 (22.01)
  Post-Treatment | 59.95 (15.74) | 60.00 (18.68)

14. Secondary Outcome: BIS/BAS Scales (Carver & White, 1994)
Description: The Behavioral Inhibition System/Behavioral Approach System Scales is a 20-item self-report where all items can be rated from 0 to 3. The total score can range from 0 to 60. Higher scores indicate higher levels of behavioral inhibition skills.
Time Frame: Measured at pre-treatment (baseline) and post-treatment (month 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unified Treatment | Wait-list Control
Number analyzed (Participants) | 26 | 11
score on a scale
  Pre-Treatment BIS | 24.15 (3.41) | 24.45 (2.16)
  Post-Treatment BIS | 22.32 (4.14) | 23.60 (2.79)
  Pre-Treatment BAS | 38.09 (6.55) | 35.18 (7.18)
  Post-Treatment BAS | 40.27 (5.78) | 35.40 (8.13)

15. Secondary Outcome: Affective Control Scale
Description: The ACS is a 42 item scale where each item is rated from 1 to 7. Scores can range from 42 to 294. Higher scores indicate higher skill levels for controlling emotions
Time Frame: Measured at pre-treatment (baseline) and post-treatment (month 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unified Treatment | Wait-list Control
Number analyzed (Participants) | 26 | 11
score on a scale
  Pre-Treatment | 140.92 (26.48) | 141.00 (35.08)
  Post-Treatment | 106.36 (25.34) | 141.60 (40.63)

16. Secondary Outcome: Anxiety Sensitivity Index
Description: The ASI is a 16 item self report where items can be scored from 0 to 4. Scores can range from 0 to 64. Higher scores indicate a higher sensitivity to anxiety and it's symptoms.
Time Frame: Measured at pre-treatment (baseline) and post-treatment (month 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unified Treatment | Wait-list Control
Number analyzed (Participants) | 26 | 11
score on a scale
  Pre-Treatment | 29.62 (11.56) | 29.27 (10.53)
  Post-Treatment | 19.36 (12.75) | 25.50 (12.40)

17. Secondary Outcome: The Thought-Action Fusion Scale (Shafran et al., 1996)
Description: The TAF is a 19 item self report where each item can be scored from 0 to 4. Scores can range from 0 to 76. Higher scores indicate a higher frequency of maladaptive cognitive intrusions.
Time Frame: Measured at pre-treatment (baseline) and post-treatment (month 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unified Treatment | Wait-list Control
Number analyzed (Participants) | 26 | 11
score on a scale
  Pre-Treatment | 13.46 (14.03) | 16.82 (15.82)
  Post-Treatment | 11.43 (9.67) | 16.90 (17.51)

18. Secondary Outcome: Intolerance of Uncertainty Scale (IUS)
Description: The IUS is a 27-item self report where each item can be scored from 0 to 4. Scores range from 0 to 108. It rates response to uncertainty, ambiguous situations, and the future. Higher scores indicate higher anxiety and depressive symptoms.
Time Frame: Measured at pre-treatment (baseline) and post-treatment (month 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unified Treatment | Wait-list Control
Number analyzed (Participants) | 26 | 11
score on a scale
  Pre-Treatment | 40.38 (20.14) | 39.27 (21.86)
  Post-Treatment | 27.77 (19.57) | 40.25 (28.38)

19. Secondary Outcome: The Trait Meta-Mood Scale (TMMS; Salovey et al., 1995)
Description: The TMMS is a 48 item self report where each item can be scored from 1 to 5. The three subscales are Attention, Clarity, and Repair. Scores for each of the three subscales can each range from 16 to 80. Higher scores indicate higher emotion regulation skills.
Time Frame: Measured at pre-treatment (baseline) and post-treatment (month 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unified Treatment | Wait-list Control
Number analyzed (Participants) | 26 | 11
score on a scale
  Pre-Treatment Attention Subscale | 76.83 (8.84) | 76.50 (9.40)
  Pre-Treatment Clarity Subscale | 50.83 (7.65) | 51.30 (11.74)
  Pre-Treatment Repair Subscale | 39.43 (4.40) | 37.40 (4.09)
  Post-Treatment Attention Subscale | 80.68 (8.12) | 76.00 (11.63)
  Post-Treatment Clarity Subscale | 54.69 (7.91) | 54.31 (11.37)
  Post-Treatment Repair Subscale | 40.59 (4.42) | 37.89 (5.53)

ADVERSE EVENTS:
Arm/Group | Unified Treatment | Wait-list Control
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/11
Other Adverse Events (participants affected / at risk) | 0/26 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes